CLINICAL TRIAL: NCT03949257
Title: Dynamic Changes of Gut Microbiota in Patients With Ulcerative Colitis After Fecal Transplantation
Brief Title: Dynamic Changes of Gut Microbiota in UC After FMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FMT-TET-190507
Record Dates: First submitted 2019-05-12; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Ulcerative Colitis
Keywords: transendoscopic enteral tubing; gut microbiota; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- colonic TET and FMT (Experimental): gut microbiota will be collected through the colonic TET after FMT
  Interventions: Device: colonic transendoscopic enteral tubing

INTERVENTIONS:
Device: colonic transendoscopic enteral tubing — Colonic transendoscopic enteral tubing (TET) is a novel, safe, convenient, and reliable way for fecal microbiota transplantation (FMT) and the whole-colon enema treatment.
  Other Names: fecal microbiota transplantation

SUMMARY:
A prospective study to investigate the dynamic changes of gut microbiota through colonic transendoscopic enteral tubing in patients with ulcerative colitis after fecal microbiota transplantation.

DETAILED DESCRIPTION:
Colonic transendoscopic enteral tubing (TET) is a novel, safe, convenient, and reliable way for fecal microbiota transplantation (FMT) and the whole-colon enema treatment. This tube also can serve as a medium for collecting gut microbiota. Fecal Microbiota Transplantation (FMT) was identified to be promising for ulcerative colitis (UC). This study aims to investigate the dynamic changes of gut microbiota in patients with UC after FMT.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed with mild or moderate ulcerative colitis.
* Patients need colonic TET and FMT
* Must be able to colonic TET and no contraindication by endoscopic examination, consent colon TET implantation and not associated with severe intestinal lesions such as fistula, stenosis, complex perianal lesions, severe ileocecal or ascending colon lesions resulting in no proper site for titanium clip fixation.
* Age > 7 years old and < 65 years old

Exclusion Criteria:

* gut microbiota was not collected successfully

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
changes of gut microbiota | 7 days
  gut microbiota will be collected through the colonic TET

SECONDARY OUTCOMES:
frequency of defecation | 7 days
  the frequency of defecation in UC patients will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: faming zhang, MD; PhD, Study Chair — The Second Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peng Z, Xiang J, He Z, Zhang T, Xu L, Cui B, Li P, Huang G, Ji G, Nie Y, Wu K, Fan D, Zhang F. Colonic transendoscopic enteral tubing: A novel way of transplanting fecal microbiota. Endosc Int Open. 2016 Jun;4(6):E610-3. doi: 10.1055/s-0042-105205. Epub 2016 Apr 28. PMID 27556065
- [Background] Westwood DA, Alexakis N, Connor SJ. Transparent cap-assisted colonoscopy versus standard adult colonoscopy: a systematic review and meta-analysis. Dis Colon Rectum. 2012 Feb;55(2):218-25. doi: 10.1097/DCR.0b013e31823461ef. PMID 22228167